CLINICAL TRIAL: NCT00288392
Title: A Double-Blind Therapeutic Exploratory Clinical Study to Evaluate the Efficacy of Soluble Beta-1,3/1,6-Glucan Compared to Placebo on Chronic Leg Ulcers in Diabetes Patients
Brief Title: Efficacy of Soluble Beta-1,3/1,6-Glucan Compared to Placebo on Chronic Leg Ulcers in Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBG-1-11
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-05

CONDITIONS: Foot Ulcer
MeSH Terms: conditions — Foot Ulcer

INTERVENTIONS:
Drug: Soluble beta-1,3/1,6-glucan

SUMMARY:
The purpose of this study is to evaluate the efficacy of soluble beta-1,3/1,6-glucan compared to placebo on the healing of chronic leg ulcers in diabetes patients.

Hypothesis: Through its ability to activate tissue macrophages and counteract diabetes-associated defects in macrophages, the soluble beta-1,3/1,6-glucan will promote the healing of leg ulcers in diabetic patients.

DETAILED DESCRIPTION:
Diabetes predisposes to ulceration of the foot through a variety of processes, including neuropathy and peripheral arterial disease. Once the skin is broken, healing is frequently delayed and the ulcer develops the biology of a chronic wound. The factors underlaying delayed healing in chronic wounds are not well understood but include the effects of repeated trauma, tissue ischemia, infection, defective white cell function, altered immune processes, and altered expression of tissue cytokines and enzymes.

Management is based on regular cleansing and debridement, off-loading and treatment of intercurrent infection with antibiotics. There are no interventions in routine use, which target aspects of chronic wound biology directly.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Age>= 18 years
* Study wound is a Wagner Grade 1 partial thickness or Grade 2 full thickness lesion but without exposed tendon, joint, or bones
* Study wound located on the foot or lower leg
* Study wound must have been present for at least 4 weeks prior to Day 0 but not longer than 2 years
* Adequate circulation to the foot, evidenced by a palpable pulse on the study foot
* Study wound > 1.0cm2 but < 20.0cm2
* Written informed consent

Exclusion Criteria:

* Pregnancy, lactation or absence of adequate contraception for fertile women
* Ankle/Brachial Index < 0.7
* Severe malnutrition
* Clinical evidence of gangrene on any part of the foot with the study wound
* Active or extensive cellulitis extending more than 1 cm beyond wound margin and/or presence of cellulitis with purulent discharge on day 0
* One or more medical condition(s) that in the opinion of the investigator would make the patient an inappropriate candidate for the study
* Active osteomyelitis of the foot with the study wound
* Necrotic toes on the foot with the study wound
* Surgical procedure (other than debridement) on the foot with the study wound the last 21 days prior to screening
* Study wound over a Charcot's joint
* Evidence of deep tissue infection of the study wound at day 0
* Non-study wound on the study foot that is located within 5.0cm from the study wound at day 0
* Random blood sugar reading > 450 mg/dL
* Alcohol or drug abuse
* Participation in other clinical studies in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06; Study Completion 2006-09

PRIMARY OUTCOMES:
- Time to healing

SECONDARY OUTCOMES:
Number of patients with complete healing of treated ulcers after 12 weeks of treatment
Percentage reduction in ulcer area of treated ulcers after 12 weeks of treatment
Percentage weekly reduction in ulcer area in treated ulcers
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Zykova, Dr.med., Principal Investigator — Municipal Healthcare Institution 1st City Hospital, Department of Endocrinology
Locations (2):
- Russia (2):
  - Municipal Healthcare Institution 1st City Clinical Hospital, Arkhangelsk
  - St. Petersburg State Institution Saint Martyr Elezabeth Hospital, Saint Petersburg

REFERENCES:
- [Derived] Zykova SN, Balandina KA, Vorokhobina NV, Kuznetsova AV, Engstad R, Zykova TA. Macrophage stimulating agent soluble yeast beta-1,3/1,6-glucan as a topical treatment of diabetic foot and leg ulcers: A randomized, double blind, placebo-controlled phase II study. J Diabetes Investig. 2014 Jul;5(4):392-9. doi: 10.1111/jdi.12165. Epub 2013 Dec 2. PMID 25411598